CLINICAL TRIAL: NCT01718990
Title: Prospective, Longitudinal Cohort Trial of Patients With Idiopathic Pulmonary Fibrosis (IPF) and Healthy Control Patients. Clinical Data, Blood, and Bronchiolavage (BAL) Fluid Will be Collected Over 12 Months.
Brief Title: Biomarker Discovery for Novel Drug Development in Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: PPG-IPF
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, Bronchiolavage (BAL) supernatant, and BAL cell pellets
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with Idiopathic Pulmonary Fibrosis (IPF): Sixty patients with IPF will be included in this prospective cohort;15 IPF patients per year for years 1-4.
- Healthy Volunteers: Sixty normal controls will be recruited from volunteers.

SUMMARY:
Drug discovery can take many years especially since most studies to measure effectiveness depend on clinical outcomes like pulmonary function tests and hospitalizations.

This is an observational study designed to collect information, blood, and bronchoalveolar lavage fluid in people who have IPF and those who do not. The people who have IPF will be followed for 12 months to collect more biological samples and record clinically relevant information.

The goal of this study is to identify new molecular markers that are measurable and reliable in people who have IPF. It is hoped that these markers can be used in future drug studies to significantly speed up the process of finding drugs that help.

ELIGIBILITY:
Inclusion Criteria:

* age 35 to 80 years
* a diagnosis of IPF by consensus criteria

Exclusion Criteria:

* any condition that makes the patient at unacceptable risk for bronchoscopy
* the presence of significant co-existing emphysema on HRCT
* active cigarette smoking (defined as smoking within the last 6 months)
* the presence of a significant co-morbidity felt to limit life expectancy to less than 12 months.
* active listing for lung transplantation
* inability to provide informed consent

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IPF
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-10; Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Molecular Markers | 12 months
  We anticipate that we will successfully enroll 60 subjects with IPF in a 12 month longitudinal cohort study and provide biological samples (Bronchiolavage (BAL), alveolar macrophages, and blood) to Projects 1-3 for use in identifying mechanistically-informative markers of alveolar epithelial cell ER stress, αvβ6-mediated TGFβ activation, and EMT. We expect that levels of some of these mechanistic markers will be measurable in patient samples, and may be differentially present in IPF compared to normal controls. Variations in baseline levels of mechanistically-informative molecular markers may identify subgroups of Idiopathic Pulmonary Fibrosis (IPF) patients that share distinct clinical phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Harold Collard, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States